CLINICAL TRIAL: NCT00361920
Title: Investigating Biomarkers of Steroid Resistant Asthma
Brief Title: Cell Biology of Steroid Resistant Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-2034
Record Dates: First submitted 2006-08-07; First posted 2006-08-09 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: steroid resistant asthma
MeSH Terms: conditions — Asthma | interventions — Prednisone

INTERVENTIONS:
Drug: prednisone

SUMMARY:
The hypothesis is that patients who demonstrate steroid resistant asthma by showing little or no improvement in lung function after a course of oral steroids have different cellular responses to steroids than patients who are steroid sensitive. These altered responses are the reason they demonstrate steroid resistance.

DETAILED DESCRIPTION:
Current NHLBI guidelines for persistent asthma management recommends the use of steroids for treatment of airway inflammation (1,2). However, some asthmatics do not respond to steroids (3-6). Unfortunately these patients are subjected to the unwanted side effects (osteoporosis, cataracts, etc) of high dose steroid therapy because non-immune tissues remain sensitive to steroids. Recent studies suggest that the costs of asthma are largely attributable to uncontrolled disease (7). Thus, it is important to understand the mechanism(s) of steroid resistance and introduce new forms of therapy for the treatment of these difficult to control asthmatics. As a prelude to pharmaceutical studies in steroid resistant asthma, it is imperative to develop biomarkers that can robustly identify individuals likely to be poor steroid responders so that alternative non-steroid anti-inflammatory therapies, such as Xolair®, can be introduced early in the course of asthma therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Will meet American Thoracic Society criteria for asthma
2. Pulmonary function tests consistent with asthma. This includes a baseline FEV1 < 80% predicted as well as a 12% improvement in FEV1 following up to 4 puffs of albuterol.
3. Subjects must be 12 to 65 years old.

Exclusion Criteria:

1. Viral infection within four weeks of the starting date.
2. Abnormal hepatic function.
3. History of COPD
4. Pregnancy.
5. History of smoking.
6. Anemia (hemoglobin less than 12 gm %)
7. Concurrent therapy with anticonvulsants, erythromycin, rifampin and any systemic asthma medication including Singular®, Xolair® or oral prednisone.
8. Greater than 500 mcg per day of inhaled corticosteroids
9. Suspected non-compliance with medical care.
10. Abnormal prednisone pharmacokinetics (applies to phase 2 of trial)
11. Patients with severe medical conditions that in the view of the investigator prohibits participation in the study (specify as required)
12. Use of any investigational agent in the last 30 days

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-08; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Assess the prevalence of steroid resistance and to determine what fraction of steroid resistant subjects have positive skin tests and IgE levels ≥30 IU/ml
Assess whether DEX-induced MKP-1 mRNA levels are decreased in PBMC or whole blood cells of SR, as compared to SS, asthmatics
Determine whether T cells from SR vs SS asthmatics proliferate in the presence of increasing concentrations of DEX
Determine whether DEX inhibits IL-6, TNF alpha, and IL-13 secretion in PBMC of SR, as compared to SS, asthmatics
Examine expression of GCR-beta and GCR alpha mRNA in PBMC of SR, as compared to SS, asthmatics, T
Analyze PBMC isolated from heparinized blood stored for 18 hours overnight at room temperature for specific aims A through D.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Leung, MD,PhD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Medical and Research Center, Denver, Colorado, United States